CLINICAL TRIAL: NCT02126462
Title: Randomized, Controlled, Phase 1 Study to Assess Safety and Immunogenicity of Co-administered Hookworm Vaccine Candidates Na-GST-1 and Na-APR-1 Adjuvanted With Alhydrogel® and Gluco-pyranosylphospho-lipid A in Gabonese Adults
Brief Title: Safety and Immunogenicity of Co-Administered Hookworm Vaccine Candidates Na-GST-1 and Na-APR-1 in Gabonese Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Maria Elena Bottazzi PhD, Sponsor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HV-001; 602843-2 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Hookworm Infection; Hookworm Disease
Keywords: Human Hookworm; Necator americanus; Hookworm; Hookworm Disease; Iron-deficiency anemia; Soil-transmitted helminth infection; Neglected Tropical Disease; Na-APR-1; Na-GST-1
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis; Anemia, Iron-Deficiency; Neglected Diseases | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 30 µg Na-GST-1 + 30 µg Na-APR-1 (M74) (Experimental): 30 µg Na-GST-1/Alhydrogel plus 5 µg GLA-AF co-administered with 30 µg Na-APR-1 (M74)/Alhydrogel plus 5 µg GLA-AF
  Interventions: Biological: Na-APR-1 (M74)/Alhydrogel®; Biological: Na-GST-1/Alhydrogel®
- Hepatitis B vaccine (Active Comparator): Hepatitis B vaccine co-administered with saline
  Interventions: Biological: Hepatitis B vaccine
- 100 µg Na-GST-1 plus 100 µg Na-APR-1 (M74) (Experimental): 100 µg Na-GST-1/Alhydrogel plus 5 µg GLA-AF co-administered with 100 µg Na-APR-1 (M74)/Alhydrogel plus 5 µg GLA-AF
  Interventions: Biological: Na-APR-1 (M74)/Alhydrogel®; Biological: Na-GST-1/Alhydrogel®

INTERVENTIONS:
Biological: Na-APR-1 (M74)/Alhydrogel®
  Arms: 100 µg Na-GST-1 plus 100 µg Na-APR-1 (M74); 30 µg Na-GST-1 + 30 µg Na-APR-1 (M74)
Biological: Na-GST-1/Alhydrogel®
  Arms: 100 µg Na-GST-1 plus 100 µg Na-APR-1 (M74); 30 µg Na-GST-1 + 30 µg Na-APR-1 (M74)
Biological: Hepatitis B vaccine — Hepatitis B vaccine co-administered with saline
  Arms: Hepatitis B vaccine

SUMMARY:
Na-GST-1 and Na-APR-1 are proteins expressed during the adult stage of the Necator americanus hookworm life cycle that are thought to play a role in the parasite's degradation of host hemoglobin for use as an energy source. Vaccination with recombinant GST-1 or APR-1 has protected dogs and hamsters from infection in challenge studies. This study will evaluate the safety and immunogenicity of co-administering Na-GST-1 and Na-APR-1 to healthy Gabonese adults living in an area of endemic hookworm infection.

DETAILED DESCRIPTION:
Double-blind, randomized, controlled dose-escalation Phase 1 clinical trial in hookworm exposed adults.

Study site: Centre de Recherches Médicales de Lambaréné Number of participants: 32 in 2 cohorts of 16

Doses of Na-GST-1 to be tested: 30 and 100 μg Doses of Na-APR-1 to be tested: 30 and 100 μg Dose of GLA-AF: 5 μg per antigen

Cohort 1: 30 μg of each of the two antigens (Na-GST-1/Alhydrogel® and Na-APR-1 (M74)/Alhydrogel®) or hepatitis B vaccine; Cohort 2: 100 μg of each of the two antigens (Na-GST- 1/Alhydrogel® and Na-APR-1 (M74) /Alhydrogel®) or hepatitis B vaccine.

Randomization: Cohort 1: 30 μg Na-GST-1 + 30 μg Na-APR-1 (M74) (n = 12) versus Hepatitis B Vaccine/placebo (n = 4) Cohort 2: 100 μg Na-GST-1 + 100 μg Na-APR-1 (M74) (n = 12) versus Hepatitis B Vaccine + placebo (n = 4)

The cohorts will be enrolled in a staggered fashion with safety data assessed prior to the Na-GST-1 and Na-APR-1 dose escalation from 30 to 100 µg.

Pre-treatment: Albendazole (400 mg) at least 2 weeks prior to first vaccination

Immunization schedule: Study days 0, 28 and 180 Route: Intramuscular in the deltoid muscle

Study duration: approximately 20 months; each participant will be followed for a total of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 50 years, inclusive, who are long-term residents of Gabon.
* Good general health as determined by means of the screening procedure.
* Assumed availability for the duration of the trial (12 months).
* Willingness to participate in the study as evidenced by signing the informed consent document.
* Negative for hookworm during screening, or if found to be infected with hookworm, has completed a course of three doses of albendazole.

Exclusion Criteria:

* Pregnancy as determined by a positive urine hCG (if female).
* Participant unwilling to use reliable contraception up until one month following the third immunization (if female and not surgically sterile, abstinent or at least 2 years post-menopausal).
* Currently lactating and breast-feeding (if female).
* Inability to correctly answer all questions on the informed consent comprehension questionnaire.
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, diabetes, or renal disease by history, physical examination, and/or laboratory studies.
* Known or suspected immunodeficiency.
* Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than 1.25-times the upper reference limit).
* Laboratory evidence of renal disease (serum creatinine greater than 1.25-times the upper reference limit, or more than trace protein or blood on urine dipstick testing).
* Laboratory evidence of hematologic disease (absolute leukocyte count <3500/mm3; absolute leukocyte count >11.0 x 103/mm3; hemoglobin <10.000 g/dl [females] or <12.0 g/dl [males]; or, platelet count <140,000/mm3).
* Other condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol.
* Participation in another investigational vaccine or drug trial within 30 days of starting this study or for the duration of the study.
* Volunteer has had medical, occupational, or family problems as a result of alcohol or illicit drug use during the past 12 months.
* History of a severe allergic reaction or anaphylaxis.
* Severe asthma as defined by the need for daily use of inhalers or emergency room/clinic visit or hospitalization within 6 months of the volunteer's planned first vaccination in the study.
* Positive for HCV
* Positive ELISA for HBsAg.
* Positive for HIV infection
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 30 days of starting this study or expect to use for the duration of the study.
* Receipt of a live vaccine within past 4 weeks or a killed vaccine within past 2 weeks prior to entry into the study.
* History of a surgical splenectomy.
* Receipt of blood products within the 6 months prior to entry into the study.
* Previous receipt of a primary series of any hepatitis B vaccine.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-11; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Vaccine-related Adverse Events | Day 360
  To estimate the frequency of vaccine-related adverse events, graded by severity, for each dose of co-administered Na-GST-1 and Na-APR-1 (M74).
  The frequency of immediate, systemic, and local injection site adverse events will be summarized. Adverse events will be assessed by study team members at 1 hour post-vaccination as well as 1, 3, 7, 14, and 28 days following each vaccination.

SECONDARY OUTCOMES:
IgG response to Na-GST-1 and Na-APR-1 (M74) | Day 194
  To determine the doses of Na-GST-1 and Na-APR-1 (M74) that generate the highest IgG antibody responses at Day 194, as determined by indirect enzyme-linked immunosorbent assays (ELISA)
Duration of antibody response to Na-GST-1 and Na-APR-1 (M74) | Day 14, 28, 42, 56, 180, 194, 208, 270, 360
  To assess and compare the duration of antibody responses to Na- GST-1 and Na-APR-1 (M74).
Exploratory studies of memory B-cell responses | Days 14, 28, 42, 56, 180, 194, 208, 270, 360
  Exploratory studies of memory B-cell responses against the metabolomics changes before and after Na-GST-1 and NA-APR-1 (M74) vaccine antigens.

CONTACTS AND LOCATIONS:
Overall Officials: Ayola Adegnika, MD, Principal Investigator — Centre de Recherches Medicales de Lambarené
Locations (1):
- Centre de Recherches Médicales de Lambaréné Albert Schweitzer Hospital, Lambaréné, Gabon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mouwenda YD, Betouke Ongwe ME, Sonnet F, Stam KA, Labuda LA, De Vries S, Grobusch MP, Zinsou FJ, Honkpehedji YJ, Dejon Agobe JC, Diemert DJ, van Leeuwen R, Bottazzi ME, Hotez PJ, Kremsner PG, Bethony JM, Jochems SP, Adegnika AA, Massinga Loembe M, Yazdanbakhsh M. Characterization of T cell responses to co-administered hookworm vaccine candidates Na-GST-1 and Na-APR-1 in healthy adults in Gabon. PLoS Negl Trop Dis. 2021 Oct 1;15(10):e0009732. doi: 10.1371/journal.pntd.0009732. eCollection 2021 Oct. PMID 34597297
- [Derived] Adegnika AA, de Vries SG, Zinsou FJ, Honkepehedji YJ, Dejon Agobe JC, Vodonou KG, Bikangui R, Bouyoukou Hounkpatin A, Bache EB, Massinga Loembe M, van Leeuwen R, Molemans M, Kremsner PG, Yazdanbakhsh M, Hotez PJ, Bottazzi ME, Li G, Bethony JM, Diemert DJ, Grobusch MP; HookVac Consortium. Safety and immunogenicity of co-administered hookworm vaccine candidates Na-GST-1 and Na-APR-1 in Gabonese adults: a randomised, controlled, double-blind, phase 1 dose-escalation trial. Lancet Infect Dis. 2021 Feb;21(2):275-285. doi: 10.1016/S1473-3099(20)30288-7. Epub 2020 Sep 11. PMID 32926834